CLINICAL TRIAL: NCT01079819
Title: Randomized, Placebo-controlled, Double-blind, Single- and Multiple-Dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of BMS-708163 in Healthy Young Male and Elderly Male and Female Chinese Subjects
Brief Title: Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of BMS-708163
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CN156-029
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2011-02-07 (Estimated); Status verified 2011-02

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — BMS 708163

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- A1 (BMS-708163) (Active Comparator)
  Interventions: Drug: BMS-708163
- A2 (Placebo) (Placebo Comparator)
  Interventions: Drug: Placebo
- B1 (BMS-708163) (Active Comparator)
  Interventions: Drug: BMS-708163
- B2 (Placebo) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMS-708163 — Capsule, Oral, 50 mg, once daily, 1 Day
  Arms: A1 (BMS-708163)
Drug: BMS-708163 — Capsule, Oral, 125 mg, once daily, 14 Days
  Arms: B1 (BMS-708163)
Drug: Placebo — Capsule, Oral, 0 mg, One daily, 1 Day
  Arms: A2 (Placebo)
Drug: Placebo — Capsule, Oral, 0 mg, One daily, 14 Day
  Arms: B2 (Placebo)

SUMMARY:
The purpose of the study is to evaluate the pharmacokinetics, safety and tolerability of BMS-708163 administered as single and multiple doses in Chinese subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects 18-45 yrs old and 65 yrs or older inclusive and postmenopausal female 65 yrs or older

Exclusion Criteria:

* Women of childbearing potential
* Gastrointestinal disorders
* Bleeding disorders
* Peptic ulcer disease
* Abnormal ECG
* Abnormal Clinical laboratory tests
* Abnormal Thyroid
* Congestive heart failure
* Cholecystectomy
* Asthma
* Hypertension
* Inability to tolerate oral medication
* Inability to be venipunctured and/or tolerate venous access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Safety assessments will be based on adverse event reports and the results of vital sign measurements, ECGs, physical exams and clinical laboratory tests. Adverse events will be tabulated and reviewed for potential significance and clinical importance | Study Day 1 through study completion + 30 days

SECONDARY OUTCOMES:
Single-dose pharmacokinetic parameters (Cmax, Tmax, AUC(0-T), AUC(INF), T-HALF and multiple-dose pk parameters (Cmax, Tmax, Cmin, AUC(TAU), T-HALF, and accumulation index will be derived from plasma concentration versus time data | Study Days 1-8 Period 1 and Days 1, 2, 5, 7, 9, 11, and 13-21 Period 2

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - West Coast Clinical Trials, Llc, Cypress, California
  - California Clinical Trials Medical Group, Glendale, California
  - Iberica Clinical Research Center, Eatontown, New Jersey

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx